CLINICAL TRIAL: NCT00187551
Title: Partial Treatment Interruptions in HIV-1 Patients With Multi-Drug Resistant Virus
Brief Title: Pilot Study Evaluating Interruption of Enfuvirtide (Fuzeon, T20) in Patients With Enfuvirtide Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Universitywide AIDS Research Program (Other)
Responsible Party: Steven Deeks, UCSF
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H8211-18804-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2006-06

CONDITIONS: HIV Infections
Keywords: enfuvirtide; T20; Fuzeon; Treatment; Interruption; Resistance; HIV Drug Resistance; Antiretroviral Agents; Salvage Therapy; Drug Resistance, Multiple; Human Immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interruption of enfuvirtide (Experimental): enfuvirtide interruption
  Interventions: Other: Interruption of enfuvirtide; Other: enfuvirtide interrupton

INTERVENTIONS:
Other: Interruption of enfuvirtide — treatment interruption
Other: enfuvirtide interrupton — enfuvitide will be interrupted in patients harboring resistant virus

SUMMARY:
The goal of this study is to examine whether enfuvirtide (T20, Fuzeon) has continued anti-HIV activity in patients experiencing an incomplete virologic response to an enfuvirtide-based regimen.

DETAILED DESCRIPTION:
Some patients do not achieve an undetectable HIV viral load with an enfuvirtide (T20, Fuzeon) based antiretroviral regimen. As a consequence, enfuvirtide resistant virus can emerge. It is not yet known if enfuvirtide has continued virologic or immunologic benefit after the drug-resistant variant emerges. Interrupting enfuvirtide may reduce the accumulation of enfuvirtide mutations and may allow for a potent response of enfuvirtide with future regimens.

Subjects must have evidence of viral replication (HIV RNA > 1,000 copies/ml on two consecutive measurements) while on a stable antiretroviral regimen containing enfuvirtide. Patients will then interrupt enfuvirtide while continuing all other antiretroviral agents. Subjects will be seen weekly for four weeks, every two weeks for an additional 8 weeks, and then every four weeks through week 48.

Plasma HIV RNA levels and CD4+/CD8+ T cell counts will be measured in real time at each visit, and provided to the referring primary care physician. Subjects will be allowed to resume enfuvirtide at any time during the course of this study. Subjects will be encouraged to resume enfuvirtide (with or without modifying the background regimen) if plasma HIV RNA levels increase by > 0.5 log on two consecutive occasions. Subjects are seen every four weeks for 24 weeks after enfuvirtide is resumed.

Plasma will be collected at those visits for HIV RNA and stored for retrospective genotype/phenotype evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving continuous enfuvirtide-based antiretroviral therapy.
* Documentation of recent plasma HIV RNA level greater than the lower limit of detection (measured within the preceding 4 weeks)
* Screening plasma HIV-1 RNA level > 1000 copies/mL.
* Negative serum pregnancy test (for women of childbearing potential) documented within the 14-day period prior to study entry.
* Subjects must be able to give written informed consent and agree to abide by the requirements of the study.

Exclusion Criteria:

* Unstable HIV disease status such that interrupting any antiretroviral therapy poses significant short-term risk for disease progression (as determined by study investigators and referring primary care provider).
* Female subjects who are pregnant, breastfeeding, or who plan to become pregnant during the study.
* Active hepatitis C infection requiring treatment with an interferon-based regimen.
* Evidence of active, untreated opportunistic infections or unexplained temperature which is > 38.5°C for seven consecutive days, within 30 days prior to the first screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
CD4 | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Deeks, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States